CLINICAL TRIAL: NCT01208571
Title: The Effect of an Interdisciplinary "Booster" Session in Primary Care Following Brief Intervention in Hospitals - a Randomized Clinical Trial
Brief Title: The Effect of a Interdisciplinary Alcohol Cessation Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-1883
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Alcohol Use Disorders
Keywords: Harmful use; Hazardous use; Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Other: "Booster session"
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: "Booster session" — Motivational interview
  Arms: Lifestyle counseling

SUMMARY:
The effect of alcohol interventions seems to be related to the intensity of the interventions. In this study the investigators will assess the effect of a interdisciplinary "booster session" in primary care, given to patients who were admitted to hospitals with alcohol related conditions, and who were given Brief Intervention before discharge. The booster session is based on a motivational interview.

DETAILED DESCRIPTION:
The study is a randomized clinical trial, and aims to recruit 60 X 2 patients. Patients admitted to Stavanger University Hospital with an alcohol contributed condition, and who has been given a brief alcohol intervention may be recruited. Candidates for secondary healthcare related to alcohol misuse will be excluded. The interdisciplinary "booster" session will be given two weeks after discharge, and will be given in the facility of the primary care physician, facilitated by both the physician and an liaison alcohol nurse from Stavanger University Hospital. The intervention is based on motivational interview technique. The primary outcome will be assessed using the Alcohol Use Disorder Identification Test-C, six months after discharge. The outcome assessor will be blinded for the intervention. All outcomes will be collected by telephone interview.

The study aims to start recruiting candidates in October-November 2010, and will stoop recruiting in December 2012 at the latest.

The study was approved by the national ethical comite in August 2011. The results of the study wil be published in international referee based journals.

ELIGIBILITY:
Inclusion Criteria:

* Admission with an alcohol related disorder

Exclusion Criteria:

* Lack of ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Disorder Identification -C (AUDIT-C) | 6 months
  Alcohol Use Disorder Identification -C. Dicothomous outcome. More or less than four points for women and five points for men.

SECONDARY OUTCOMES:
Timeline followback | 6 months
  Grams og alcohol pr week.
Readmissions | 6 months
  Readmission to a hospital for an alcohol related and/or a non-alcohol related condition within six months after discharge.
Readiness to Change Questionaire (RTCQ) | 6 months
  Continous variable
Quality of Life | 6 months
  SF 12

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Oppedal, MD, Study Chair — Helse Stavanger HF; Sverre Nesvaag, Dr, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway